CLINICAL TRIAL: NCT01325818
Title: The Effects of Pravastatin and Rosuvastatin on the Tissue Characteristics and Morphology of Coronary Plaques in Patients With Stable Angina Pectoris
Brief Title: The Effects of Pravastatin and Rosuvastatin on Coronary Plaques in Patients With Stable Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Yokohama City University Medical Center, Cardiovascular Center, Yokohama City University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YCUMC20110324
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Disease; Hypercholesterolemia
Keywords: Coronary Artery Disease; Coronary Disease; Dyslipidemia; Stable Angina Pectoris; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases Pravastatin; Rosuvastatin; Anticholesteremic Agents; Antilipemic Agents; Antimetabolites; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Therapeutic Uses; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: conditions — Coronary Disease; Hypercholesterolemia; Coronary Artery Disease; Dyslipidemias; Angina, Stable; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases | interventions — Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1:pravastatin, 2:rosuvastatin (Active Comparator): 1. Active Comparator Drug:pravastatin
  2. Active Comparator Drug:rosuvastatin
  Interventions: Drug: pravastatin, rosuvastatin

INTERVENTIONS:
Drug: pravastatin, rosuvastatin — 1. Active Comparator Intervention: Drug: pravastatin 10mg/day or 20mg/day
  2. Active Comparator Intervention: Drug: rosuvastatin 20mg/day

SUMMARY:
The purpose of this study is to compare the effects of pravastatin and rosuvastatin on coronary plaque characteristics in patients with stable angina pectoris.

DETAILED DESCRIPTION:
Previous mega trials have demonstrated that lipid-lowering therapy with HMG-CoA reductase inhibitors in individuals with high risk of cardiovascular disease reduces the incidence of coronary heart disease. NCEP ATP-III has suggested the advantage of more intensive lipid lowering therapy with a goal of reducing LDL-C below 70 mg/dL for such patients categorized as very high risk. In Japan, Japan Atherosclerosis Society (JAS) Guidelines for Diagnosis and Treatment of Atherosclerotic Cardiovascular Diseases 2002 have recommended that an LDL-C goal for patients with coronary heart disease (CHD) should be below 100 mg/dL. However, there is no satisfactory evidence whether the investigators need to lower LDL-C level less than the 70mg/dL or not in Japanese population.

Recently, research on diagnosis of coronary plaque has shown significant advances. The REVERSAL study in patients with a history of CHD, by diagnosis with intravascular ultrasound (IVUS), suggested that intensive lipid lowering therapy with atorvastatin (80 mg/day) was associated with no growth of plaque (-0.4% compared to baseline), whereas therapy with pravastatin (40 mg/day) showed a slight increase (2.7%) in plaque volume over 18 months in Western population.

MEGA study has shown that lipid lowering therapy with pravastatin (10-20 mg/day) was associated with a 33% reduction in coronary heart disease incidence as the primary prevention in Japanese patients. However, the effect of lipid lowering therapy in secondary prevention of cardiovascular events is unknown.

Relative plaque regression rate between intensive and moderate lipid lowering therapy would clarify the ideal level of target LDL-C in Japanese population. Furthermore, the different effect on coronary plaque between pravastatin and rosuvastatin which have different LDL-C lowering effect and different affinity to arterial tissue would determine the superior lipid lowering regimen to affect coronary plaque volume.

Therefore, the aim of the present study is to evaluate whether there would be lipid lowering therapy differences in terms of the composition of coronary artery plaques in patients with stable angina pectoris (SAP) using integrated backscatter intravascular ultrasound (IB-IVUS) and optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed as stable angina pectoris, and successful percutaneous coronary intervention (PCI) were performed with intravascular ultrasound (IVUS) and optical coherence tomography (OCT) guidance.
2. Patients having coronary plaques (≧ 500 µm in thickness or % plaque of 20% or more at ≧ 5 mm distal or proximal to the previously treated area in the same branch of coronary artery.
3. Patients with dyslipidemia as defined by any of the following criteria:

   * TC ≧ 220 mg/dL
   * LDL-C ≧ 140 mg/dL
   * Cholesterol-lowering treatment is allowed according to the investigator's judgment when LDL-C ≧ 100 mg/dL or TC ≧ 180mg/dL.
   * Patients who are under cholesterol-lowering treatment and LDL-C ≦ 120 mg/dL
4. Patients 20 years or older at the time of their consent.
5. Patients with written consent by their own volition after being provided sufficient explanation for their participation in this clinical trial.

Exclusion Criteria:

1. Patients with bypass graft or in-stent restenosis at the site of PCI.
2. Patients who received PCI in the past on the lesion where the evaluation of coronary plaque volume is planned.
3. Patients who had plaques in a non-culprit site and might receive PCI during the treatment period.
4. Patients receiving lipid-lowering drugs (fibrates, probucol, nicotinic acid, cholestyramine or cholesterol absorption inhibitors).
5. Patients with familial hypercholesterolemia.
6. Patients with cardiogenic shock.
7. Patients receiving cyclosporine.
8. Patients with any allergy to pravastatin and rosuvastatin.
9. Patients with hepatobiliary disorders.
10. Pregnant women, women suspected of being pregnant, or lactating women.
11. Patients with renal disorders (Cr≧2.0mg/dL) or undergoing dialysis.
12. Patients who are ineligible in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-03 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
the percent change in fibrous cap thickness by optical coherence tomography | 9-11 months
  the percent change in fibrous cap thickness by optical coherence tomography

SECONDARY OUTCOMES:
the percent change and the absolute change from baseline in coronary plaque volume and IB signal obtained by IB-IVUS | 9-11 months
  the percent change and the absolute change from baseline in coronary plaque volume, the percent change in integrated backscatter signal obtained by integrated backscatter IVUS
the absolute change from baseline in number of TCFA and plaque rupture, and in neointima thickness on stent struts by OCT | 9-11 months
  the absolute change from baseline in number of TCFA, plaque rupture, thrombus, calcification, and in neointima thickness on stent struts by optical coherence tomography
the percent change and the absolute change from baseline in total cholesterol and LDL cholesterol | 9-11 months
  the percent change and the absolute change from baseline in total cholesterol and low-density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hibi, Study Chair — Yokohama City University Medical Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Japan